CLINICAL TRIAL: NCT02079194
Title: Comparison Between P2Y12 Antagonist MonotHerapy and Dual Antiplatelet Therapy in Patients UndergOing Implantation of Coronary Drug-Eluting Stents
Brief Title: Comparison Between P2Y12 Antagonist Monotherapy and Dual Antiplatelet Therapy After DES
Acronym: SMART-CHOICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Hyeon-Cheol Gwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMC 2014-01-161
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Coronary Artery Disease
Keywords: Drug-eluting stents; aspirin; P2Y12 antagonist monotherapy
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- P2Y12 antagonist monotherapy (Experimental): P2Y12 antagonist monotherapy after 3-month DAPT
  Interventions: Drug: P2Y12 antagonist monotherapy
- Aspirin + P2Y12 antagonist (Experimental): Aspirin + P2Y12 antagonist after 3-month DAPT
  Interventions: Drug: aspirin plus P2Y12 antagonist

INTERVENTIONS:
Drug: P2Y12 antagonist monotherapy
  Arms: P2Y12 antagonist monotherapy
Drug: aspirin plus P2Y12 antagonist
  Arms: Aspirin + P2Y12 antagonist

SUMMARY:
To compare the efficacy and safety of clopidogrel monotherapy versus aspirin plus P2Y12 antagonist following 3-month of DAPT in patients undergoing PCI with DES.

DETAILED DESCRIPTION:
This trial is a prospective, randomized, multi-center, open label, noninferiority trial. Patients undergoing PCI with DES will be eligible. After successful PCI with DES, all eligible patients will be randomized either to clopidogrel monotherapy or to aspirin plus P2Y12 antagonist following 3-month of DAPT.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 20 years of age.
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.
* Patients undergoing successful PCI

Exclusion Criteria:

* Hemodynamic instability or cardiogenic shock
* Active bleeding
* Known hypersensitivity or contraindication to study medications
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study
* Non-cardiac co-morbid conditions are present with life expectancy <2 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* DES implantation within 12 months before index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2014-03-18 (Actual); Primary Completion 2018-07-07 (Actual); Study Completion 2020-07-07 (Estimated)

PRIMARY OUTCOMES:
A composite of death, myocardial infarction, or cerebrovascular events | 1 year
  12 months after the index procedure

SECONDARY OUTCOMES:
All cause Death | 1 years
cardiac death | 1 years
Myocardial infarction (MI) | 1 years
Cerebrovascular accident (CVA) | 1 years
Target lesion revascularization (TLR) | 1 years
Target vessel revascularization (TVR) | 1 years
Any revascularization | 1 years
Stent thrombosis: definite or probable stent thrombosis by ARC definition | 1 years
BARC bleeding ≥2 | 1 years
BARC bleeding ≥3 | 1 years
Major adverse cardiocerebral event (MACCE): death, MI, CVA, or any revascularization | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Hyeon-Cheol Gwon, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Cardiac and Vascular Center; Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Song PS, Seong SW, Kim JY, An SY, Kim MJ, Ahn KT, Jin SA, Jeong JO, Yang JH, Hahn JY, Gwon HC, Jang WJ, Yoon HJ, Bae JW, Choi WG, Song YB. The Association of CHADS-P2A2RC Risk Score With Clinical Outcomes in Patients Taking P2Y12 Inhibitor Monotherapy After 3 Months of Dual Antiplatelet Therapy Following Percutaneous Coronary Intervention. Korean Circ J. 2024 Apr;54(4):189-200. doi: 10.4070/kcj.2023.0268. PMID 38654565
- [Derived] Shin ES, Her AY, Kim B, Hahn JY, Song YB, Lee JM, Park TK, Yang JH, Choi JH, Choi SH, Lee SH, Gwon HC; SMART-CHOICE Investigators. Sex-Based Outcomes of P2Y12 Inhibitor Monotherapy After Three Months of Dual Antiplatelet Therapy in Patients Undergoing Percutaneous Coronary Intervention. J Korean Med Sci. 2023 Nov 20;38(45):e383. doi: 10.3346/jkms.2023.38.e383. PMID 37987108
- [Derived] Choi KH, Park YH, Song YB, Park TK, Lee JM, Yang JH, Choi JH, Choi SH, Oh JH, Chun WJ, Jang WJ, Im ES, Jeong JO, Cho BR, Oh SK, Yun KH, Cho DK, Lee JY, Koh YY, Bae JW, Choi JW, Lee WS, Yoon HJ, Lee SU, Cho JH, Choi WG, Rha SW, Gwon HC, Hahn JY; SMART-CHOICE Investigators. Long-term Effects of P2Y12 Inhibitor Monotherapy After Percutaneous Coronary Intervention: 3-Year Follow-up of the SMART-CHOICE Randomized Clinical Trial. JAMA Cardiol. 2022 Nov 1;7(11):1100-1108. doi: 10.1001/jamacardio.2022.3203. PMID 36169938
- [Derived] Lee SH, Lee SY, Chun WJ, Song YB, Choi SH, Jeong JO, Oh SK, Yun KH, Koh YY, Bae JW, Choi JW, Gwon HC, Hahn JY. Clopidogrel monotherapy in patients with and without on-treatment high platelet reactivity: a SMART-CHOICE substudy. EuroIntervention. 2021 Dec 3;17(11):e888-e897. doi: 10.4244/EIJ-D-21-00223. PMID 34031020
- [Derived] Song PS, Park YH, Oh JH, Song YB, Choi SH, Gwon HC, Cho DK, Rha SW, Bae JW, Jeong JO, Hahn JY; SMART-DATE and the SMART-CHOICE investigators. P2Y12 Inhibitor Monotherapy Versus Conventional Dual Antiplatelet Therapy or Aspirin Monotherapy in Acute Coronary Syndrome: A Pooled Analysis of the SMART-DATE and SMART-CHOICE Trials. Am J Cardiol. 2021 Jul 1;150:47-54. doi: 10.1016/j.amjcard.2021.03.053. Epub 2021 May 16. PMID 34011436
- [Derived] Kim J, Jang WJ, Lee WS, Choi KH, Lee JM, Park TK, Yang JH, Choi JH, Song YB, Choi SH, Gwon HC, Lee SH, Oh JH, Chun WJ, Park YH, Im ES, Jeong JO, Cho BR, Oh SK, Yun KH, Cho DK, Lee JY, Koh YY, Bae JW, Choi JW, Yoon HJ, Lee SU, Cho JH, Choi WG, Rha SW, Hahn JY. P2Y12 inhibitor monotherapy after coronary stenting according to type of P2Y12 inhibitor. Heart. 2021 Jun 11;107(13):1077-1083. doi: 10.1136/heartjnl-2020-318821. PMID 33758008
- [Derived] Yun KH, Lee SY, Cho BR, Jang WJ, Song YB, Oh JH, Chun WJ, Park YH, Im ES, Jeong JO, Oh SK, Cho DK, Lee JY, Koh YY, Bae JW, Choi JW, Lee WS, Yoon HJ, Lee SU, Cho JH, Choi WG, Rha SW, Lee JM, Park TK, Yang JH, Choi JH, Choi SH, Lee SH, Gwon HC, Hahn JY; SMART-CHOICE Investigators [Link]. Safety of 3-Month Dual Antiplatelet Therapy After Implantation of Ultrathin Sirolimus-Eluting Stents With Biodegradable Polymer (Orsiro): Results From the SMART-CHOICE Trial. J Am Heart Assoc. 2021 Jan 5;10(1):e018366. doi: 10.1161/JAHA.120.018366. Epub 2020 Dec 21. PMID 33345567
- [Derived] Hahn JY, Song YB, Oh JH, Chun WJ, Park YH, Jang WJ, Im ES, Jeong JO, Cho BR, Oh SK, Yun KH, Cho DK, Lee JY, Koh YY, Bae JW, Choi JW, Lee WS, Yoon HJ, Lee SU, Cho JH, Choi WG, Rha SW, Lee JM, Park TK, Yang JH, Choi JH, Choi SH, Lee SH, Gwon HC; SMART-CHOICE Investigators. Effect of P2Y12 Inhibitor Monotherapy vs Dual Antiplatelet Therapy on Cardiovascular Events in Patients Undergoing Percutaneous Coronary Intervention: The SMART-CHOICE Randomized Clinical Trial. JAMA. 2019 Jun 25;321(24):2428-2437. doi: 10.1001/jama.2019.8146. PMID 31237645
- [Derived] Song YB, Oh SK, Oh JH, Im ES, Cho DK, Cho BR, Lee JY, Lee JM, Park TK, Yang JH, Choi JH, Choi SH, Lee SH, Gwon HC, Hahn JY. Rationale and design of the comparison between a P2Y12 inhibitor monotherapy versus dual antiplatelet therapy in patients undergoing implantation of coronary drug-eluting stents (SMART-CHOICE): A prospective multicenter randomized trial. Am Heart J. 2018 Mar;197:77-84. doi: 10.1016/j.ahj.2017.12.002. Epub 2017 Dec 6. PMID 29447787